CLINICAL TRIAL: NCT04802148
Title: Alveolar Ridge Preservation in Molar Extraction Sockets With an Open Healed Collagen Membrane: A Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202004006RINB
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-04

CONDITIONS: Tooth Extraction
Keywords: ridge preservation, tooth extraction, collagen membrane, cone-beam computed tomography
MeSH Terms: interventions — Punctal Plugs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (natural healing) (No Intervention): Extraction socket is naturally healed
- Test 1 (membrane guided regeneration) (Experimental): Extraction socket is filled with graft (FDBA) and covered with collagen membrane
  Interventions: Procedure: membrane guided regeneration
- Test 2 (collagen plug) (Active Comparator): Extraction socket is filled with a collagen plug
  Interventions: Procedure: collagen plug

INTERVENTIONS:
Procedure: membrane guided regeneration — after tooth extraction, the socket was filled with membrane and graft (FDBA)
  Arms: Test 1 (membrane guided regeneration)
Procedure: collagen plug — after tooth extraction, the socket was filled with collagen plug
  Arms: Test 2 (collagen plug)

SUMMARY:
The resorption of alveolar ridge after tooth extraction develop difficulty in restoring the extraction area with implant or bridge. Therefore, try to preserve the alveolar ridge width and height at extraction socket and gaining its bone volume in maximal is worth for clinical investigation. There are several method to deal with alveolar ridge preservation (ARP), the most popular way for its approach, the trend is toward to minimally invasive treatment. Alveolar ridge preservation which is done with open-healed wound without primary closure is the key for minimally invasive approach.

This three-armed randomized clinical trial would like to determine the effect of applying ribose cross-linked collagen membrane without primary flap closure in molar extraction sockets for alveolar ridge preservation. The procedure is for implant site development.

Three groups were designed as test group1 was grafted with freeze dried bone allograft (FDBA) and covered by ribose cross-linked collagen membrane (OSSIX® PLUS). In test group2 sockets filled with collagen plug(Teruplug®) and sockets healed naturally as control group. Cone-beam computed tomography(CBCT) scans are obtained immediately and 4 months after ARP as the primary outcome and secondary outcome. A biopsy from implant site and histomorphometric analysis will be done as well. The change of marginal bone level and the width/height of keratinized mucosa are measured.

ELIGIBILITY:
Inclusion Criteria:

* Age>20
* according to periapical film, the bone defect over bucco-lingual and mesio-distal direction less than 50%
* patient agreed to undergo implant therapy after tooth extraction

Exclusion Criteria:

* systemic diseases which will affect wound healing (ex. Diebetes)
* heavy smoker (10 cigarette/day)
* patient who underwent oral-maxillary surgery or who diagnosed with oral cancer
* patient who is pregnant or who is breast-feeding
* patient who is allergic to Lidocaine
* patient who cannot cooperate the study design

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
alveolar ridge width and height in three plane | four months after surgery
  mesure with CBCT

SECONDARY OUTCOMES:
gingival thickness | four months after surgery
  measure with CBCT and clinical observation

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No